CLINICAL TRIAL: NCT02331212
Title: Role of Hyaluronic Acid in Cancer Stem Cell Niche
Brief Title: Role of Hyaluronic Acid in Causing Cancer Stem Cell Growth in the Bones of Patients With Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Logistical Issues
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00030529; NCI-2014-02554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 74A14; CCCWFU 74A14; CCCWFU 74A14 (Other: Wake Forest University Health Sciences); R01CA173499 (NIH); P30CA012197 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2015-01-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Breast Carcinoma Metastatic to the Bone; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (role of HAS2+ in CSCs): Blood and bone marrow samples are collected and analyzed via flow cytometry and PCR. Cells are also transplanted into mice and studied.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies the role of a substance called hyaluronic acid in causing the growth of cancer stem cells in the bones of patients with breast cancer. Cancer stem cells are a type of cancer cells that may cause the cancer to spread to other parts of the body. Studying samples of blood and bone marrow from patients and animal models in the laboratory may help doctors learn more about whether hyaluronic acid affects the growth of cancer in the bones.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the hypothesis that there are more hyaluronan synthase 2 (HAS2)+ cells in patients with bone metastasis compared to patients with only local disease.

SECONDARY OBJECTIVES:

I. To evaluate the hypothesis that cells with HAS2+ and cancer stem cell (CSC)+ (cluster of differentiation [CD]24-/CD44+/epithelial specific antigen [ESA]+) cells will have the most aggressive growth in the bone, using an animal model.

OUTLINE:

Blood and bone marrow samples are collected and analyzed via flow cytometry and polymerase chain reaction (PCR). Cells are also transplanted into mice and studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, histologically confirmed primary and/or metastatic breast cancer
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with newly diagnosed, histologically confirmed primary and/or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
HAS2 expression, measured by single-cell PCR | Baseline
  Descriptive statistics will be generated. The relationship of each cell's bone metastatic ability and HAS2 expression will be examined using correlations within each group between these two measures. The mean values of the HAS2 expression and bone metastatic ability will be compared between groups using one-way analysis of variance (ANOVA) models. In addition, 2-sample t-tests will be used to compare the primary cancer and bone metastases groups.

SECONDARY OUTCOMES:
CSC marker expression | Baseline
  Expression of CSC markers including CD24, CD44 and ESA will be examined. These will also be examined using descriptive statistics and compared with each other using one-way ANOVA models and 2-sample t-tests to compare the primary cancer and bone metastases groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kounosuke Watabe, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States